CLINICAL TRIAL: NCT01740128
Title: A Hebbian Approach to Regaining Control of Spared Circuits in Spinal Cord Injury
Brief Title: Multimodal Exercises to Improve Leg Function After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B0881-W; 5IK2RX000881-03 (NIH); 01407 (Other: Bronx VA Medical Center); SPU-11-077 (Other: Bronx VA Medical Center)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Spinal Cord Injuries; Paraplegia; Paraparesis
Keywords: spinal cord injuries; paraplegia; postural balance; locomotor activity; exercise therapy; electromyography; transcranial magnetic stimulation, single pulse
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Paraparesis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Multimodal then Treadmill training (Experimental): Participants will undergo harness-supported multimodal balance training exercises while simultaneously performing skilled hand exercises. Following a washout period of at least 6 weeks, Participants will undergo body weight supported treadmill training using the Lokomat apparatus.
  Interventions: Device: Robotic body weight supported treadmill training; Other: Harness-supported multimodal balance training
- Treadmill then Multimodal training (Active Comparator): Robotic body weight supported treadmill training will be applied using the Lokomat apparatus. Following a washout period of at least 6 weeks, Participants will undergo harness-supported balance training exercises while simultaneously performing skilled hand exercises.
  Interventions: Device: Robotic body weight supported treadmill training; Other: Harness-supported multimodal balance training

INTERVENTIONS:
Device: Robotic body weight supported treadmill training — 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
  Other Names: Lokomat
Other: Harness-supported multimodal balance training — 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
  Other Names: balance exercises, skilled hand exercises

SUMMARY:
Many people with spinal cord injury (SCI) retain at least some movement below their injury, but their muscles often have a 'mind of their own'. Typical exercise programs focus on keeping muscles strong and flexible, but don't usually focus on helping patients control their muscles. The investigators' exercise research study will compare two different programs with the specific goal of improving conscious control of patients' muscles below the injury. This study focuses on those with 'chronic' SCI - the injury occurred at least one year prior to enrolling.

This is a single center study taking place in the Bronx, NY.

The first phase of the study will be observational - the investigators will analyze which nerve connections might remain partially intact through the injury (even if the nerves aren't consciously controlled). Participants with all severity of SCI may participate in this first phase.

The second phase of the study will involve people who retain at least slight ability to move their legs and the ability to move the arms against gravity. Each person will undergo two different exercise rehabilitation strategies: weight-supported treadmill training; and balance training combined with skilled arm or hand exercises.

The investigators will compare the effects of these exercise programs on a variety of outcomes, including gait speed, balance, strength, and muscle activation in response to brain stimulation.

The investigators hypothesize that participants with chronic SCI undergoing combined balance/arm/hand training will show improved outcomes when compared to traditional gait or balance training.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 21-65 years;
* SCI duration > 12 months;
* SCI level C2-T12;
* All SCI severity eligible for baseline testing;
* For exercise protocol, must have severity of Grade C or D on American Spinal Injury Association (ASIA) Impairment Scale, or volitional strength of at least 1/5 in two or more key lower extremity muscles, as well as at least 3/5 in both shoulder and elbow muscles;
* Able to tolerate upright position with support;
* Morphologically capable of fitting a weight-support harness and robotic treadmill system;
* Ability to give informed consent.

Exclusion Criteria:

* Unsuitable cognitive capacity as judged by the study physician;
* Diagnosis of neurological injury other than SCI, such as stroke, traumatic brain injury, or other neurological condition that the study physician considers to be exclusionary;
* Multiple spinal cord lesions;
* History of frequent autonomic dysreflexia;
* History of seizures;
* Use of medications that significantly lower seizure threshold, such as anti-psychotics, tricyclic antidepressants, amphetamines, and bupropion;
* History of implanted brain/spine/nerve stimulators, aneurysm clips, or cardiac pacemaker/defibrillator;
* Deep vein thrombosis in lower extremities of less than 6 months duration;
* Pregnancy;
* (Interventional phase only): Lack of detectable tibialis anterior motor evoked potential (MEP) at baseline even with active facilitation;
* (Interventional phase only): Pressure ulcers greater than stage 1 severity on the foot, ankle, knee and/or pelvic girdle;
* (Interventional phase only): Bone mineral density of the hip (proximal femur) T-score <3.5 standard deviations from age- and gender-matched normative data;
* (Interventional phase only): Any spasticity, contractures, or heterotopic ossification that result in inadequate range of motion of the shoulder, elbow, wrist, fingers, hip, knee, or ankle joints in the judgment of the study physician;
* (Interventional phase only): Inability to cooperate with instructions or unwilling to commit to daily training sessions for 3-4 days per week over 12-16 weeks;
* (Interventional phase only): A diagnosis of coronary artery disease that precludes moderate to intense exercise.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y Harel, MD PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.

REFERENCES:
- [Background] Harel NY, Asselin PK, Fineberg DB, Pisano TJ, Bauman WA, Spungen AM. Adaptation of computerized posturography to assess seated balance in persons with spinal cord injury. J Spinal Cord Med. 2013 Mar;36(2):127-33. doi: 10.1179/2045772312Y.0000000053. PMID 23809527
- [Background] Harel NY, Martinez SA, Knezevic S, Asselin PK, Spungen AM. Acute changes in soleus H-reflex facilitation and central motor conduction after targeted physical exercises. J Electromyogr Kinesiol. 2015 Jun;25(3):438-43. doi: 10.1016/j.jelekin.2015.02.009. Epub 2015 Mar 2. PMID 25771437

RESULTS

PARTICIPANT FLOW:
Groups:
- Multimodal Then Treadmill Training: Participants will undergo harness-supported multimodal balance training exercises while simultaneously performing skilled hand exercises. Following a washout period of at least 6 weeks, Participants will undergo body weight supported treadmill training using the Lokomat apparatus.
  Multimodal training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
- Treadmill Then Multimodal Training: Participants will undergo body weight supported treadmill training using the Lokomat apparatus. Following a washout period of at least 6 weeks, Participants will undergo harness-supported multimodal balance training exercises while simultaneously performing skilled hand exercises.
  Robotic body weight supported treadmill training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
Period: Overall Study
Arm/Group | Multimodal Then Treadmill Training | Treadmill Then Multimodal Training
Started | 10 | 11
Completed | 4 | 4
Not Completed | 6 | 7
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Insufficient protocol compliance | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Multimodal Then Treadmill Training: Participants will undergo harness-supported multimodal balance training exercises while simultaneously performing skilled hand exercises. Following a washout period of at least 6 weeks, Participants will undergo body weight supported treadmill training using the Lokomat apparatus.
  Multimodal training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
  Robotic body weight supported treadmill training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
- Treadmill Then Multimodal Training: Robotic body weight supported treadmill training will be applied using the Lokomat apparatus. Following a washout period of at least 6 weeks, Participants will undergo harness-supported balance training exercises while simultaneously performing skilled hand exercises.
  Multimodal training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
  Robotic body weight supported treadmill training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Multimodal Then Treadmill Training | Treadmill Then Multimodal Training | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Evoked Potential (MEP) Amplitude in the Tibialis Anterior Muscle at the End of Training.
Description: Change between baseline and Evaluation #2 in motor evoked potential area in the tibialis anterior muscle.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Only two participants in the study had consistent MEPs at baseline.
Measure: Number; unit: Amplitude percentage of Mmax
Groups:
- Multimodal Training: Participants will undergo harness-supported balance training exercises while simultaneously performing skilled hand exercises.
  Multimodal training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
- Treadmill Training: Robotic body weight supported treadmill training will be applied using the Lokomat apparatus.
  Robotic body weight supported treadmill training: 30-minute sessions will be conducted 3-4 times per week for a total of 48 sessions over 12 to 16 weeks.
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 1 | 1
Amplitude percentage of Mmax | -1.75 | -2.01

2. Secondary Outcome: Change From Baseline in ISNCSCI Lower Extremity Motor Score.
Description: Change between baseline and Evaluation #2 in lower extremity motor score derived from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI). Range of scores 0-50, higher is better.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: One subject in multimodal group failed to appear for post-intervention testing for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 9 | 10
units on a scale | 0.11 (4.81) | -0.30 (4.32)

3. Secondary Outcome: Change From Baseline in Berg Balance Scale Sitting With Back Unsupported Score.
Description: Change between baseline and Evaluation #2 in Berg sitting unsupported subscore. Range 0-4, higher better.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Incomplete analysis due to dropouts before post-testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 10 | 8
units on a scale | 0.10 (0.32) | 0.00 (0.00)

4. Secondary Outcome: Change in Leg Spasticity on Modified Ashworth Scale
Description: Change between baseline and Evaluation #2 in modified Ashworth Scale. 0-4 score, lower is better.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Incomplete analysis due to dropouts before post-testing, and due to incomplete outcome assessment by Investigating team.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 4 | 9
units on a scale | 0.13 (0.25) | -0.39 (0.89)

5. Secondary Outcome: Change in Gait Speed on 10-meter Walk Test.
Description: Change between baseline and Evaluation #2 in gait speed during 10-meter walk test.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Insufficient number of participants able to walk at baseline.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 1 | 3
meters per second | .04 (0) | 0.12 (0.132)

6. Secondary Outcome: Change From Baseline in Walking Index for Spinal Cord Injury II (WISCI II) Scale.
Description: Change between baseline and Evaluation #2 in WISCI II score. Scores range 0-20, higher is better.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Insufficient number of participants able to walk at baseline. Measure not recorded by Investigating team.
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Total Number of Steps Taken by Both Feet During Seated 10-second Step Test.
Description: Change between baseline and Evaluation #2 in steps taken during 10-second step test.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Low number of participants able to perform seated steps at baseline.
Measure: Mean (Standard Error); unit: steps
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 4 | 4
steps | 2.83 (1.14) | -1.08 (1.03)

8. Secondary Outcome: Change in Subjective Pain as Determined by McGill Pain Questionnaire (Short Form).
Description: Change between baseline and Evaluation #2 in McGill Pain Questionnaire (Subjective Domain). Total scale 0-45, lower is better.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Incomplete analysis due to dropouts before post-testing, and due to incomplete outcome assessment by Investigating team.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 9 | 7
units on a scale | 0.89 (2.76) | -0.93 (3.00)

9. Secondary Outcome: Change From Baseline in Endpoint Excursion and Directional Control Parameters Achieved During Seated Limits of Stability Testing.
Description: Seated posturography performed using the "Limits of Stability" module of the Smart EquiTest apparatus (Neurocom) while seated. Directional Control measure.
Time Frame: Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Incomplete analysis due to dropouts before post-testing.
Measure: Mean (Standard Error); unit: Percentage of perfect path to target
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 10 | 9
Percentage of perfect path to target | 1.93 (3.42) | 8.42 (4.02)

10. Secondary Outcome: Change From Baseline in Soleus H-reflex Facilitation.
Description: Change between baseline and Evaluation #2 in soleus H-reflex facilitation by transcranial magnetic stimulation (TMS). Short-interval 0-20ms.
Time Frame: Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Incomplete analysis due to dropouts before post-testing, and due to lack of soleus H-reflex in several subjects.
Measure: Mean (Standard Error); unit: percentage of control reflex size
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 7 | 8
percentage of control reflex size | 6.63 (6.25) | -5.20 (3.35)

11. Secondary Outcome: Changes From Baseline in Survey: Spinal Cord Injury - Spasticity Evaluation Tool (SCI-SET)
Description: Change between baseline and Evaluation #2 in SCI-SET score. Range of scores -105 to +105. Higher is better.
Time Frame: Eval #1 at baseline; Eval #2 at end of training (48 sessions, average 3-4 months)
Population: Incomplete analysis due to dropouts before post-testing, and due to incomplete outcome assessment by Investigating team.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multimodal Training | Treadmill Training
Number analyzed (Participants) | 7 | 6
units on a scale | 2.14 (11.44) | -0.67 (0.82)

ADVERSE EVENTS:
Time Frame: Approx. 6 months or until completion of study participation.
Description: No serious adverse events. Several minor skin abrasions.
Arm/Group | Multimodal Training | Treadmill Training
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Multimodal Training (N=10) | Treadmill Training (N=11)
skin abrasion (Skin and subcutaneous tissue disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Smaller than expected enrollment, high dropout rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes